CLINICAL TRIAL: NCT06877533
Title: A First-in-Human Open-label, Phase I/Ib Dose Escalation and Expansion Cohort Study of EOS006215 as Monotherapy and in Combination With Pembrolizumab or Other Anticancer Treatments in Participants With Advanced Solid Tumors
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The study was terminated early due to sponsor's strategic business decision.
Sponsor: iTeos Belgium SA (Industry)
Responsible Party: Sponsor
Organization: iTeos Therapeutics (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TRM-010; 2024-520369-30-00 (EU CTIS Number)
Record Dates: First submitted 2025-03-10; First posted 2025-03-14 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-08

CONDITIONS: Selected Advanced Solid Tumors
Keywords: Advanced solid tumors; Cancer; Phase I; Immunotherapy; Anticancer; Anti-PD1; TREM2; Pembrolizumab; EOS-215; Metastatic; Antibodies; Monoclonal antibodies; Antineoplastic therapy; EOS006215
MeSH Terms: conditions — Neoplasms; Neoplasm Metastasis | interventions — Antineoplastic Agents

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Part 1 Dose Escalation (Monotherapy) (Experimental): EOS006215 dose escalation as monotherapy
  Interventions: Drug: EOS006215
- Part 1 Dose Escalation (Combination Therapy) (Experimental): EOS006215 dose escalation in combination with pembrolizumab or with other anticancer agents
  Interventions: Drug: EOS006215; Drug: Anticancer agent

INTERVENTIONS:
Drug: EOS006215 — Multiple doses of EOS006215
Drug: Anticancer agent — Multiple doses of EOS006215 in combination with other anticancer agents
  Arms: Part 1 Dose Escalation (Combination Therapy)

SUMMARY:
TRM-010 is a first-in-human (FIH) clinical study designed to assess the safety, tolerability, pharmacokinetics (PK), pharmacodynamics (PD), and preliminary antitumor activity of EOS006215, a fully human monoclonal antibody that binds to the triggering receptor expressed on myeloid cells 2 (TREM2). The study includes EOS006215 monotherapy and combination therapy with other anticancer agents in participants with advanced solid tumors.

DETAILED DESCRIPTION:
The study will be conducted in 2 parts:

* Part 1 - Dose Escalation Phase I dose escalation cohorts for EOS006215 as monotherapy and in combination with anticancer treatments in participants with specific tumor types.
* Part 2 - Dose Expansion Phase Ib dose expansion cohort(s) may be included to further evaluate the safety, tolerability, efficacy, PK and PD of EOS006215 as monotherapy or in combination with anticancer treatments in participants with specific tumor types.

ELIGIBILITY:
Inclusion Criteria:

* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Histologically or cytologically confirmed advanced or metastatic unresectable solid tumors for which standard approved treatment is not available or the participant is ineligible or did not tolerate the standard approved treatment.
* At least one tumor lesion measurable per RECIST v1.1
* Have an estimated minimum life expectancy of ≥ 12 weeks.
* Adequate organ/marrow and liver function
* Agree to use adequate highly effective method of contraception during the study is mandatory, if WOCBP or male

Exclusion Criteria:

* Prior systemic anticancer treatment including investigational agents within 3 weeks (or 5 half-lives, whichever is shorter) before the first dose of study treatment
* Major surgery planned or within 5 weeks before the first dose of study treatment, or minor surgical procedure (except tumor biopsy) within 7 days before the first dose of study treatment.
* Radiotherapy within 2 weeks before the first dose of study treatment.
* Evidence of severe active or chronic infections requiring systemic antibacterial, antiviral, or antifungal treatment, including tuberculosis infection
* Known seropositivity for or active infection with human immunodeficiency virus (HIV)
* Known seropositivity for hepatitis B virus (HBV), with evidence of active HBV infection
* Known seropositivity for hepatitis C virus (HCV), with evidence of active HCV infection
* Live or live-attenuated vaccine within 30 days before the first dose of study treatment.
* History or current evidence of uncontrolled or significant cardiovascular disease
* History or current evidence of significant autoimmune disease that required systemic
* treatment
* Diagnosis of immunodeficiency or any condition requiring systemic treatment with immunosuppressive medication
* Pregnant or breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2025-04-07 (Actual); Primary Completion 2025-07-10 (Actual); Study Completion 2025-07-10 (Actual)

PRIMARY OUTCOMES:
Incidence of dose-limiting toxicities (DLTs), adverse events (AEs)/serious adverse events (SAEs) [Safety and Tolerability] | DLTs - At the end of Cycle 1 AEs/SAES - Duration of intervention (up to 24 months) plus 30 days follow-up
Rate of treatment modifications (interruption or permanent discontinuation) [Safety and Tolerability] | Duration of intervention (up to 24 months)
Changes in safety parameters (clinical laboratory tests, vital signs, and electrocardiogram [ECG] / QTcF) [Safety and Tolerability] | Duration of intervention (up to 24 months) plus 30 days follow-up

SECONDARY OUTCOMES:
Overall response rate (ORR) [Efficacy] | From randomization to confirmed radiological improvement, if applicable, assessed up to 24 months.
  Proportion of participants with Best Overall Response (BOR) of complete response (CR) or partial response (PR) confirmed at a minimum of 2 post-baseline radiological assessments, without an intervening response of progressive disease
Duration of response (DoR) | From first confirmed CR or PR (whichever is first recorded) until the date of documented disease progression or death in the absence of disease progression, assessed up to 24 months.
  Time from the date of first confirmed CR or PR (whichever is first recorded) until the date of documented disease progression or death in the absence of disease progression.
Progression-free survival (PFS) per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 [Efficacy] | Time from starting treatment until disease progression or death for any reason.
Serum concentrations and PK parameters of EOS006215 | From start of treatment until end of treatment (EOT)
  Serum concentration-time data will be summarized by descriptive statistics by each treatment cohort and time point. PK parameters, such as Cmax, Cmin, AUC and CL will be derived by non-compartmental analysis and summarized with descriptive statistics.
Incidence of antidrug antibody (ADA) against EOS006215 | From start of treatment until end of treatment (EOT)
  Individual ADA occurrence will be listed, and percentage of occurrence will be summarized by descriptive statistics.
Dose-finding to determine recommended Phase 2 dose | Duration of intervention (up to 24 months) plus 30 days follow-up
  The RP2D(s) will be identified from the available safety, tolerability, PK, PD and preliminary efficacy data across the dose ranges evaluated in monotherapy and in combination with anticancer agents.

CONTACTS AND LOCATIONS:
Overall Officials: iTeos Belgium SA, Study Director — iTeos Belgium SA
Locations (2):
- United States (2):
  - Sarah Cannon Research Institute at HealthOne, Denver, Colorado
  - Florida Cancer Specialists (FSC SAC DDU) Sarasota, Sarasota, Florida

IPD SHARING:
Plan to Share IPD: No